CLINICAL TRIAL: NCT05076227
Title: Comparison of Different BNT162b2 and ChAdOx1-S COVID-19 Vaccination Intervals and Combinations on Reactogenicity and Humoral Immunogenicity in Adults
Brief Title: Effect of Different SARS-CoV-2 Vaccine Schedules and Vaccination Intervals on Reactogenicity and Humoral Immunogenicity
Status: Completed | Type: Observational
Sponsor: Serge Thal (Other)
Responsible Party: Sponsor-Investigator, Serge Thal, Clinical Professor, Head of anaesthesiology, University of Witten/Herdecke
Organization: University of Witten/Herdecke (Other)
Other Study IDs: HelCoVac
Record Dates: First submitted 2021-02-23; First posted 2021-10-13 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: SARS-CoV2 Infection; Immunisation Reaction; Antibody Hypersensitivity; Tolerance
Keywords: SARS-CoV2; COVID-19; mRNA vaccination; vector based vaccination; heterlogues vaccination; homologues vaccination; HelCoVac; Helios Hildesheim COVID-19 Vaccination Study
MeSH Terms: conditions — COVID-19 | interventions — ChAdOx1 nCoV-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- BNT162b2/BNT162b2 - 3 wks: hospital staff receiving BioNTech as prime vaccination and also receiving BioNTech after 3 weeks as boost vaccination
  Interventions: Drug: IM injection of vaccination (mRNA vaccination)
- ChAdOx1/ChAdOx1 - 12 wks: hospital staff receiving AstraZeneca as prime vaccination and also receiving AstraZeneca as boost vaccination after 12 weeks
  Interventions: Drug: IM injection of vaccination (vector based vaccination)
- ChAdOx1/BNT162b2 - 12 wks: hospital staff receiving AstraZeneca as prime vaccination and receiving BioNTech as boost vaccination after 12 weeks
  Interventions: Drug: IM injection of vaccination (mRNA vaccination); Drug: IM injection of vaccination (vector based vaccination)
- BNT162b2/BNT162b2 - 6 wks: hospital staff receiving BioNTech as prime vaccination and also receiving BioNTech after 6 weeks as boost vaccination
  Interventions: Drug: IM injection of vaccination (mRNA vaccination)

INTERVENTIONS:
Drug: IM injection of vaccination (mRNA vaccination) — mRNA vaccination
  Other Names: Cormirnaty (BioNTech/Pfizer)
  Groups: BNT162b2/BNT162b2 - 3 wks; BNT162b2/BNT162b2 - 6 wks; ChAdOx1/BNT162b2 - 12 wks
Drug: IM injection of vaccination (vector based vaccination) — vector based vaccination
  Other Names: AZD1222 (AstraZeneca)
  Groups: ChAdOx1/BNT162b2 - 12 wks; ChAdOx1/ChAdOx1 - 12 wks

SUMMARY:
Investigation of the reactogenicity and immunogenicity of homologous and heterologous vaccine combinations with regard to the formation of SARS-CoV-2 antispike antibodies in health care workers after basic immunization and boost vaccination

DETAILED DESCRIPTION:
The basic immunizations (first and second vaccination) were performed from January to June 2021 using the m-RNA vaccine BNT162b2 (BioNTech/Pfizer, B)9 and the vector-based vaccine ChAdOx1-S (AstraZeneca, A). BNT162b2 was used to boost vaccine all study population. The time interval between the basic immunisation and the boost vaccination varied.

Four vaccine-groups could be distinguished:

Group 1 received BNT162b2 with the second vaccination 3 weeks after the first vaccination.

Vaccinees of groups 2 and 3 received AZD1222/ChAdOx1-S as first vaccination and could choose after 12 weeks whether second vaccination with BNT162b2 or AZD1222/ChAdOx1-S should be carried out. This results in homologous (first: AZD1222/ChAdOx1-S, second: AZD1222/ChAdOx1-S) and heterologous (first: AZD1222/ChAdOx1-S, second: BNT162b2) vaccine combinations.

Group 4 received BNT162b2 with the second vaccination 6 weeks after first vaccination.

Blood samples were collected at six time points: four weeks, three and six months after completion of the basic immunization, immediately before boost vaccination, four weeks and three months after boost vaccination.

Reactogenicity after first, second, and boost vaccination was assessed using questionnaires to determine vaccine-induced adverse drug reactions (ADR) within seven days after the respective vaccinations.

In addition, demographic data (age, gender, occupational group, allergies) were collected, local and systemic vaccination reactions are differentiated and the need for medication and inability to work as a result of vaccination reactions are prospectively recorded.

ELIGIBILITY:
Inclusion Criteria:

* hospital staff who received COVID-19 vaccination

Exclusion Criteria:

* lack of a written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hospital staff willing to be vaccinated against SARS-Cov-2 (COVID-19)
Sampling Method: Non-Probability Sample
Enrollment: 1206 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2022-03-27 (Actual); Study Completion 2022-03-27 (Actual)

PRIMARY OUTCOMES:
Difference between the four cohorts regarding the antibody of the viral spike protein 4 weeks after second vaccination | 4 weeks after second vaccination
  The descriptive data are described by frequencies (%/n) and the continuous data by corresponding position parameters (median, interquartile range). The confirmatory analysis is performed using the Wilcoxon or Kruskal-Wallis test.
  The Bonferroni correction is applied accordingly.
Difference between the four cohorts regarding the antibody of the viral spike protein 3 months after second vaccination | 3 months after second vaccination
  The descriptive data are described by frequencies (%/n) and the continuous data by corresponding position parameters (median, interquartile range). The confirmatory analysis is performed using the Wilcoxon or Kruskal-Wallis test.
  The Bonferroni correction is applied accordingly.
Difference between the four cohorts regarding the antibody of the viral spike protein 6 months after second vaccination | 6 months after second vaccination
  The descriptive data are described by frequencies (%/n) and the continuous data by corresponding position parameters (median, interquartile range). The confirmatory analysis is performed using the Wilcoxon or Kruskal-Wallis test.
  The Bonferroni correction is applied accordingly.
Difference between the four cohorts regarding the antibody of the viral spike protein directly before boost vaccination | directly before boost vaccination
  The descriptive data are described by frequencies (%/n) and the continuous data by corresponding position parameters (median, interquartile range). The confirmatory analysis is performed using the Wilcoxon or Kruskal-Wallis test.
  The Bonferroni correction is applied accordingly.
Difference between the four cohorts regarding the antibody of the viral spike protein 4 weeks after boost vaccination | 4 weeks after boost vaccination
  The descriptive data are described by frequencies (%/n) and the continuous data by corresponding position parameters (median, interquartile range). The confirmatory analysis is performed using the Wilcoxon or Kruskal-Wallis test.
  The Bonferroni correction is applied accordingly.
Difference between the four cohorts regarding the antibody of the viral spike protein 3 months after boost vaccination | 3 months after boost vaccination
  The descriptive data are described by frequencies (%/n) and the continuous data by corresponding position parameters (median, interquartile range). The confirmatory analysis is performed using the Wilcoxon or Kruskal-Wallis test.
  The Bonferroni correction is applied accordingly.

SECONDARY OUTCOMES:
Do the four cohorts differ in terms of reactogenicity (systemic and/or local vaccine reactions) after the first vaccination? | immediately after first vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Do the four cohorts differ in terms of reactogenicity (systemic and/or local vaccine reactions) after the second vaccination? | immediately after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Do the four cohorts differ in terms of reactogenicity (systemic and/or local vaccine reactions) after the boost vaccination? | immediately after third (boost) vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Differences between the 4 groups after first vaccination regarding a. the individual local vaccination reactions? b. the individual systemic vaccination reactions? c. the number or percentage of vaccination reactions? | immediately after first vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Differences between the 4 groups after second vaccination regarding a. the individual local vaccination reactions? b. the individual systemic vaccination reactions? c. the number or percentage of vaccination reactions? | immediately after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Differences between the 4 groups after boost vaccination regarding a. the individual local vaccination reactions? b. the individual systemic vaccination reactions? c. the number or percentage of vaccination reactions? | immediately after boost vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Is there a difference between the four cohorts regarding the severity of vaccination reactions? | immediately after first vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Is there a difference between the four cohorts regarding the severity of vaccination reactions? | immediately after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Is there a difference between the four cohorts regarding the severity of vaccination reactions? | immediately after boost vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Do the four cohorts differ with respect to the temporal occurrence of vaccination reactions? | immediately after first vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Do the four cohorts differ with respect to the temporal occurrence of vaccination reactions? | immediately after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Is there a difference between the four cohorts regarding the use of medication due to vaccination reactions? | first and second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Do the four cohorts differ with regard to the need for a certificate of incapacity for work due to vaccination reactions? | immediately after first vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Are there differences regarding the job groups and the vaccination week days? | immediately after first vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Do the four cohorts differ with regard to the need for a certificate of incapacity for work due to vaccination reactions? | immediately after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Are there differences regarding the job groups and the vaccination week days? | immediately after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Do the four cohorts differ with regard to the need for a certificate of incapacity for work due to vaccination reactions? | immediately after boost vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Are there differences regarding the job groups and the vaccination week days? | immediately after boost vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Are there differences within the cohorts regarding vaccination reactions in subjects with a known allergy? | immediately after first vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Are there differences within the total population regarding vaccination reactions in subjects with a known allergy? | immediately after first vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Are there differences within the cohorts regarding vaccination reactions in subjects with a known allergy? | immediately after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Are there differences within the total population regarding vaccination reactions in subjects with a known allergy? | immediately after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Is there a correlation within cohorts or within the overall population at four weeks regarding the level of antibody and the a. Extent of vaccine response (local, systemic, local & systemic, none)? b. Gender? c. Age? d. BMI? | 4 weeks after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. Spearman's correlation is calculated.
Do the variables listed above have an influence on the level of antibody? | 4 weeks after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. To investigate a potential influence of the variables, a logistic regression is performed if necessary.
Is there a correlation within cohorts or within the overall population at 3 months regarding the level of antibody and the a. Extent of vaccine response (local, systemic, local & systemic, none)? b. Gender? c. Age? d. BMI? | 3 months after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. Spearman's correlation is calculated.
Do the variables listed above have an influence on the level of antibody? | 3 months after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. To investigate a potential influence of the variables, a logistic regression is performed if necessary.
Is there a correlation within cohorts or within the overall population at 6 months regarding the level of antibody and the a. Extent of vaccine response (local, systemic, local & systemic, none)? b. Gender? c. Age? d. BMI? | 6 months after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. Spearman's correlation is calculated.
Do the variables listed above have an influence on the level of antibody? | 6 months after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. To investigate a potential influence of the variables, a logistic regression is performed if necessary.
Is there a correlation within cohorts or within the overall population directly before the boost regarding the level of antibody and the a. Extent of vaccine response (local, systemic, local & systemic, none)? b. Gender? c. Age? d. BMI? | directly before boost vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively.
Do the variables listed above have an influence on the level of antibody? | directly before boost vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively.
Is there a correlation within cohorts or within the overall population at 4 weeks after boost regarding the level of antibody and the a. Extent of vaccine response (local, systemic, local & systemic, none)? b. Gender? c. Age? d. BMI? | 4 weeks after boost vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively.
Do the variables listed above have an influence on the level of antibody? | 4 weeks after boost vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively.
Is there a correlation within cohorts or within the overall population at 3 months after boost regarding the level of antibody and the a. Extent of vaccine response (local, systemic, local & systemic, none)? b. Gender? c. Age? d. BMI? | 3 months after boost vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively.
Do the variables listed above have an influence on the level of antibody? | 3 months after boost vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively.
Is there a statistically significant or clinically relevant difference between the (drop in) antibodies at three months from baseline within the four cohorts? | 3 months after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Is there a statistically significant or clinically relevant difference between the (drop in) antibodies at six months from baseline within the four cohorts? | 6 months after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Is there a statistically significant or clinically relevant difference between the (drop in) antibodies at three months from baseline between the four cohorts? | 3 months after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Is there a statistically significant or clinically relevant difference between the (drop in) antibodies at six months from baseline between the four cohorts? | 6 months after second vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Are there any subjects within the study follow-up period who had proven SARS Cov2 infection? (Comparison between groups) | until end of study
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively. The analysis is performed using appropriate tests such as Fisher's exact test, Chi² test, Mann-Whitney U test or Kruskal-Wallis test.
Is there a correlation within the overall population between the level of antibody and detected SARS Cov2 infection? | 3 months and 6 months after second vaccination, directly before boost vaccination and 4 weeks and 3 months after boost vaccination
  For the secondary endpoints, frequencies (%/n) for categorical data and corresponding measures of location (median, interquartile range) for continuous data are used descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Serge C Thal, MD, Study Chair — University of Witten/Herdecke; Michael Dedroogh, MD, Principal Investigator — Helios Clinical Hildesheim
Locations (1):
- Helios Hospital Hildesheim, Hildesheim, Lower Saxony, Germany